CLINICAL TRIAL: NCT06681142
Title: Pharmacist-physiotherapist Collaborative Management for Early Knee Osteoarthritis
Acronym: PACE-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00145908
Record Dates: First submitted 2024-11-03; First posted 2024-11-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis (OA) of the Knee; Physiotherapy; Pharmacy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Control) Group (No Intervention): Pharmacists will provide a general educational pamphlet and will inform the primary care physician of patient participation and referral for further assessment of knee OA.
  Participants randomized to this group will be offered physiotherapy and/or pharmacy interventions (individual or GLA:D program 3 months after enrollment) and pharmacy options (comprehensive medication review). It will be explained to participants that usual care is 'conservative therapy'.
  Usual care participants will be eligible to opt in for a comprehensive medication review (pharmacist) and/or the physiotherapy sessions and will be evaluated at 9-months after enrollment.
- Intervention Group (Experimental): Pharmacists will provide comprehensive 1:1 patient care, including a SCHOLAR assessment and medication review, provide specific drug therapy recommendation(s) using shared decision making (SDM), and provide comprehensive patient education/resources. Pharmacists will refer to physiotherapy clinics located nearby for patient convenience and to establish community pharmacy/physiotherapy clinic relationships.
  Participants will be offered a physiotherapy assessment at a nearby physiotherapy clinic within 2 weeks of being assessed by the pharmacist. After the physiotherapy assessment session, participants who are diagnosed with symptomatic knee OA will be offered 1) up to 5 individual physiotherapy sessions within a 6-week period, or 2) the GLA:D program for knee OA which includes 6-weeks of neuromuscular exercises along with 2 education session in a group format.
  Interventions: Other: Pharmacy-Physiotherapy Intervention

INTERVENTIONS:
Other: Pharmacy-Physiotherapy Intervention — Pharmacists will provide comprehensive 1:1 patient care, including a complete patient assessment and medication review, provide specific drug therapy recommendation(s) using shared decision making (SDM), and provide patient education, including further written materials.
  Participants will be offered either individual or group physiotherapy sessions at the a private clinic.
  Arms: Intervention Group

SUMMARY:
Osteoarthritis (OA) is a slowly progressive chronic condition that is associated with aging and is characterized as joint pain. Individuals with early-stage OA usually do not seek medical attention. If and when they do, patients more often present to a pharmacy for over-the-counter medications.

The investigators want to leverage community pharmacists' accessibility and scope of practice to best support patients with early knee OA. Given there are no disease-modifying treatments for OA, treatment guidelines center on patient education, self-management, and exercise, with medications playing a supporting role. Self-management is an effective strategy that provides a solid foundation for managing this progressive chronic condition and health care professionals like physiotherapists and pharmacists can help with the development and application of these skills.

DETAILED DESCRIPTION:
Pharmacists will identify patients with knee pain using two recruitment strategies: (1) Posters placed near the dispensary and 'shelf talkers' placed near the over-the-counter non- steroidal anti-inflammatory drugs, acetaminophen, and natural health products (e.g. glucosamine, collagen) will recommend patients with knee pain talk to their pharmacist and (2) Patients receiving care by a pharmacist for other conditions that have similar risk factors as OA will be asked about symptomatic knee OA (e.g. obesity).

The inclusion criteria is patients 50 years of age or older who have been regularly experiencing pain, aching, or stiffness in and/or around the knee for at least 1 month. The exclusion criteria is patients with prior knee surgery, history of acute knee injury (6 months), unable or unwilling to attend physiotherapy, previous physician diagnoses of inflammatory arthritis or fibromyalgia, and unable to speak/ read English.

For those patients with probable symptomatic knee OA, the study will be explained and upon agreement, written consent will be secured. Following enrollment, the pharmacist will ask participants to complete the baseline assessments (in pharmacy or online):

* Knee injury and OA Outcome Score (KOOS) -Reason for visiting the pharmacy
* Socio-demographics (DOB, sex/gender, education, marital status, employment) -Past medical history (chronic conditions, current medications, height/weight, other joint involvement) -Previous medications/injections trialed for knee pain -Lifestyle activities (smoking, alcohol use, walking tolerance and any assistive walking devices) -Co-interventions (eg. chiropractor, joint injections, naturopath) -Self-management (Patient Activation Measure) The pharmacist will also answer questions that participants may have regarding services and medications.

Participants will be randomized to either the control arm which is usual care or the intervention arm which includes a referral to physiotherapy and a comprehensive medication review. Randomization will occur in variable computer-generated blocks of 4-8 participants. Following the enrolment, the pharmacist will receive a code that randomizes the patients into either the treatment group (comprehensive pharmacist assessment, pharmacologic recommendations, and education with referral to physiotherapy) or usual care (brief assessment and recommendation by the pharmacist, education information brochure).

If participants have a family physician, the pharmacist will provide a notice that the patient likely has knee OA and is enrolled in this study. The name of the pharmacist and physiotherapist will be provided.

ELIGIBILITY:
Inclusion Criteria:

* regularly experiencing pain, aching, or stiffness in and/or around the knee for at least 1 month
* complete the screening PhIT-OA questionnaire

Exclusion Criteria:

* prior knee surgery
* history of acute knee injury (6 months)
* unable or unwilling to attend physiotherapy
* previous physician diagnoses of inflammatory arthritis or fibromyalgia
* unable to speak/ read English

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Disease specific self-report measure for OA | Baseline, Post Intervention (3 & 6 month after baseline)
  The Knee Injury in OA Outcome Score (KOOS) from 0-100 where a higher score is a better outcome.

SECONDARY OUTCOMES:
Patient Activation Measure (PAM) | Baseline, Post Intervention (3 & 6 month after baseline)
  Scale from 0-100 where a higher score is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, Principal Investigator — University of Alberta; Jill Hall, Principal Investigator — University of Alberta; Allyson Jones, Principal Investigator — University of Alberta
Locations (1):
- Mint Health & Drugs Festival Place Sherwood Park, Sherwood Park, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided